CLINICAL TRIAL: NCT06637358
Title: A Text-based Reduction Intervention for Smokeless Tobacco Cessation- Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00103410 _1
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Smokeless Tobacco Cessation
Keywords: Smokeless Tobacco; Quitting Smokeless Tobacco; Quit Coach
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended Scheduled Gradual Reduction (SGR) (Active Comparator): Extended scheduled gradual reduction. Participants are asked to gradually reduce smokeless tobacco usage.
  Interventions: Behavioral: Extended Scheduled Gradual Reduction (SGR)
- Quit Coach and Extended Scheduled Gradual Reduction (SGR) (Experimental): Extended scheduled gradual reduction given with the extra support of a live text-based coach. Participants are asked to gradually reduce smokeless tobacco usage and engage in weekly check-ins with their assigned quit coach.
  Interventions: Behavioral: Extended Scheduled Gradual Reduction (SGR); Behavioral: Quit Coach

INTERVENTIONS:
Behavioral: Extended Scheduled Gradual Reduction (SGR) — The extended SGR program will allow participants additional time to reduce smokeless tobacco use until they reach zero. The intent of this program is to reduce the number of times participants use smokeless tobacco down to zero. Participants will also receive text-based support messages.
Behavioral: Quit Coach — Weekly check-ins and support will be given to this group via the quit coach interactions. The intent of this program is to reduce the number of times participants use smokeless tobacco down to zero. Participants will also receive text-based support messages.
  Arms: Quit Coach and Extended Scheduled Gradual Reduction (SGR)

SUMMARY:
All participants will receive the EnufSnuff.TXT scheduled gradual reduction (SGR) intervention for 6 weeks and, for those who do not reach the point of quit, includes getting randomized (like the flip of a coin) into either an additional 8-10 weeks of the EnufSnuff.TXT intervention or into receiving an additional 8-10 weeks of the EnufSnuff.TXT intervention along with a dedicated text quit coach to send and receive live support.

DETAILED DESCRIPTION:
All participants will receive the EnufSnuff.TXT intervention (a text-based personalized reduction plan and daily text-based cessation support messages) for 6 weeks and, for those who report that they have not achieved complete cessation, includes getting randomized into either an additional 8-10 weeks of the EnufSnuff.TXT intervention or into receiving an additional 8-10 weeks of the EnufSnuff.TXT intervention along with a dedicated quit coach to send and receive live text support. The investigators will conduct phone-based or smart phone-based assessments with participants at baseline, end of program, and 7-month follow-up after intervention completion. The investigators will also conduct a brief midpoint check (after the first 6 weeks of intervention) with participants to ask if they have quit using smokeless tobacco. Research staff will email participants redcap surveys at baseline, end of program, and 7-months. Participants will be able to opt for a recorded telephone interview at the 7-month check-in. Each opted-in participant will be interviewed only once.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older
2. Have used smokeless tobacco for the last year, currently dip 3 or more times a day
3. Have an address in a rural census tract defined by a RUCC code of 4-10 and/or an IMU of 62 or lower
4. Interested in participating in a cessation program; and
5. Have access to a cell phone with unlimited texting ability.

Exclusion Criteria:

1. Non-English speaking;
2. Have smoked cigarettes or used any other tobacco product in the past 30 days (i.e., dual user) and are not willing to abstain during the intervention period
3. Currently participating in a smokeless tobacco cessation study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-11-04 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by the number of recruited individuals who enrolled | Baseline
Feasibility as measured by the number of participants who left the study (attrition) | Up to 6 months
Acceptability as measured by the number of participants who found the intervention useful | Up to 6 months
  As measured via telephone interview.
Acceptability as measured by the number of participants who reported that the intervention received changed their smokeless tobacco use | Up to 6 months
  As measured via telephone interview.
Acceptability as measured by the number of participants who reported that the intervention made them think about quitting | Up to 6 months
  As measured via telephone interview.
Acceptability as measured by the number of participants who reported that they would recommend the program to a friend | Up to 6 months
  As measured via telephone interview.
Preliminary efficacy as measured by the number of participants who quit smokeless tobacco by the end of treatment | Up to approximately 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Devon Noonan, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-04-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT06637358/ICF_000.pdf